CLINICAL TRIAL: NCT03508960
Title: The Chinese Early-onset Parkinson's Disease Registry
Brief Title: Chinese EOPD Registry
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CEOPDR
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — extraction of DNA from peripheral blood

SUMMARY:
The purpose of the Chinese Early-onst Parkinson's disease Registry (CEOPDR) is to develop a database of persons with early-onset Parkinson's disease (EOPD) in China.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common disorder among degenerative neurological disease. Early-onset PD (EOPD) has its unique clinical feature and genetic basis.Investigators aim to establish a database of EOPD,and characterize the clinical feature, genetic basis, environmental factors and their interactions EOPD in China.

Method:

1. Clinical feature will be measured by scales and neurological tests.Standard scales includes: Unified Parkinson's Disease Rating Scale(UPDRS), Hoehn-Yahr stages, NMSS, MMSE, PDSS(Parkinson disease sleep scales),Rapid Eye Movement Sleep Behaviour Disorder Questionnaire(RBDQ-HK),ESS(Epworth Sleepiness Scale),Rome III functional constipation scale，SCOPA-AUT (the Scale for Outcomes in PD for Autonomic Symptoms)，PFS(Parkinson Fatigue Scale)，CH-RLSq，Hyposmia rating scale(HRS)HAMILT depression scale，the 39-item Parkinson's Disease Questionnaire(PDQ-39)，Freezing of gait scale(FOG)，dyskinesia related scales, Wearing-off scale(WO)
2. Peripheral blood from patients was collected for whole exome sequencing.
3. The environmental factors are explored by questionnaires including smoking,drinking, pesticide and heavy metals.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD by UKBB and other standard criteria Age of onset is no more than 50 years old.

Exclusion Criteria:

* Patients have a family history of PD.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: PD patients with early-onset
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Database of Early-onset Parkinson's Disease | 10 years
  To collect 3000 patients with early-onset parkinson's disease and establish the database of early-onset Parkinson's disease in mainland China.
Risk Factors | 10 years
  To characterize clinical feature and environmental factors among Chinese early-onset parkinson's disease
Genetic Basis | 10 years
  To characterize the genetic basis of Chinese EOPD and detect clinically relevant genetic variants in these cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Yang Y, Tang BS, Weng L, Li N, Shen L, Wang J, Zuo CT, Yan XX, Xia K, Guo JF. Genetic Identification Is Critical for the Diagnosis of Parkinsonism: A Chinese Pedigree with Early Onset of Parkinsonism. PLoS One. 2015 Aug 21;10(8):e0136245. doi: 10.1371/journal.pone.0136245. eCollection 2015. PMID 26295349
- [Background] Liu ZH, Guo JF, Li K, Wang YQ, Kang JF, Wei Y, Sun QY, Xu Q, Wang DL, Xia K, Yan XX, Xu CS, Tang BS. Analysis of several loci from genome-wide association studies in Parkinson's disease in mainland China. Neurosci Lett. 2015 Feb 5;587:68-71. doi: 10.1016/j.neulet.2014.12.027. Epub 2014 Dec 17. PMID 25528405
- [Background] Li K, Tang BS, Liu ZH, Kang JF, Zhang Y, Shen L, Li N, Yan XX, Xia K, Guo JF. LRRK2 A419V variant is a risk factor for Parkinson's disease in Asian population. Neurobiol Aging. 2015 Oct;36(10):2908.e11-5. doi: 10.1016/j.neurobiolaging.2015.07.012. Epub 2015 Jul 11. PMID 26234753
- [Result] Liu Z, Tang B, Guo J, Zhou X, Sun Q, Xu Q, Xu C, Yan X. Mutations analysis of RAB39B gene in Chinese early-onset Parkinson's disease. Parkinsonism Relat Disord. 2016 Jul;28:157-8. doi: 10.1016/j.parkreldis.2016.03.019. Epub 2016 Mar 24. No abstract available. PMID 27036214
- [Result] Fan K, Tang BS, Wang YQ, Kang JF, Li K, Liu ZH, Sun QY, Xu Q, Yan XX, Guo JF. The GBA, DYRK1A and MS4A6A polymorphisms influence the age at onset of Chinese Parkinson patients. Neurosci Lett. 2016 May 16;621:133-136. doi: 10.1016/j.neulet.2016.04.014. Epub 2016 Apr 13. PMID 27085534